CLINICAL TRIAL: NCT01762163
Title: Efficacy and Safety of Qizhitongluo Capsule in the Recovery Phase of Ischemic Stroke With Qi Deficiency and Blood Stasis Syndrome: a Multicenter, Randomized,Double-blind，Placebo- and Active-controlled Adaptive Study
Brief Title: Efficacy and Safety of Qizhitongluo Capsule in the Recovery Phase of Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QZTL2013; QZTL (Registry Identifier: QZTL)
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke,adaptive design, randomized, double-blind
MeSH Terms: conditions — Ischemic Stroke | interventions — naoxintong

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Qizhitongluo Capsule (Experimental): Basic treatment：Aspirin Enteric-coated Tablets was administered orally at a dosage of 100mg/d once per night;the routine recovery training.
  intervention treatment:the Capsules were administered orally, four capsules each time, three times a day after each meal（placebo was taken only after lunch, and Qizhitongluo Capsule was taken after breakfast and supper)for 12 weeks.
  Interventions: Drug: Qizhitongluo Capsule; Drug: Aspirin Enteric-coated Tablets; Behavioral: the routine recovery training; Drug: placebo
- Naoxintong Capsule (Active Comparator): Basic treatment：Aspirin Enteric-coated Tablets was administered orally at a dosage of 100mg/d once per night; the routine recovery training.
  intervention treatment:Naoxintong Capsule was administered orally, four capsules each time, three times a day after each meal for 12 weeks.
  Interventions: Drug: Naoxintong Capsule; Drug: Aspirin Enteric-coated Tablets; Behavioral: the routine recovery training
- Placebo (Placebo Comparator): Basic treatment：Aspirin Enteric-coated Tablets was administered orally at a dosage of 100mg/d once per night and the routine recovery training.
  intervention treatment:placebo capsule was administered orally four capsules each time, three times a day after each meal for 12 weeks.
  Interventions: Drug: Aspirin Enteric-coated Tablets; Behavioral: the routine recovery training; Drug: placebo

INTERVENTIONS:
Drug: Qizhitongluo Capsule
  Other Names: QZTL group
  Arms: Qizhitongluo Capsule
Drug: Naoxintong Capsule
  Other Names: NXT group
  Arms: Naoxintong Capsule
Drug: Aspirin Enteric-coated Tablets
Behavioral: the routine recovery training
Drug: placebo
  Arms: Placebo; Qizhitongluo Capsule

SUMMARY:
This is a 20-week study consisting of a 12-week multicenter, randomized,double-blind adaptive study to compare efficacy and safety of Qizhitongluo Capsule,Naoxintong Capsule and placebo in the recovery phase of ischemic stroke with qi deficiency and blood stasis syndrome, and a 8-week post-treatment safety follow-up.After 312 patients complete 12 weeks of treatment there will be an interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age≥35 years and <80 years;
* Diagnosis of ischemic stroke in recovery phase, according to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2010;
* Diagnosis of ischemic stroke with qi deficiency and blood stasis syndrome;
* The interval from the onset to recruitment was 15-28 days;
* FM score <90 or AQ<93.8 and diagnosis of aphasia;
* Diagnosis of cerebral anterior circulation obstruction;
* 4≤ NIHSS score<20;
* Patient is willing to participate voluntarily and to sign a written patient informed consent.

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) or other cerebral diseases (eg.vascular malformation, tumor, abscess or multiple sclerosis etc.) on CT or MRI.
* Known history of allergy or suspected allergic to the study drugs.
* Liver function impairment with the value of ALT or AST over 1.5-fold of normal value.
* Renal dysfunction with the value of serum creatinine over 1.5-fold of normal value.
* Cerebral embolism caused by cerebral tumor, cerebral trauma, cerebral parasitosis, rheumatic heart disease, coronary heart disease or other cardiac diseases complicated with atrial fibrillation.
* Prestroke score on the mRS ≥2.
* Space-occupying lesions, CT or MRI revealed midline structure shift; CT revealed that massive cerebral infarction including more than one lobe of brain or over 1/3 of blood-supply area of middle cerebral artery.
* Disable patients prescribed by law（blind, deaf, dumb, mental retardation, mental disorders and physical disabilities which due to other causes affect neural function deficient scale).
* Hemorrhagic tendency or recent severe or dangerous bleeding in 3 months.
* Suspected addicted into alcohol or drug abuse; with severe complications that would make the condition more complicated assessed by the investigator.
* Woman with pregnancy, lactation or positive result of pregnancy test, or women who want to be pregnant in recent.
* Patient who is participating in other trials or has been participated in other trials in recent 3 months.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in the Lower Extremity Fugl-Meyer score | baseline, after 4,12 weeks of treatment, after 90 days of onset.

SECONDARY OUTCOMES:
Change in Aphasia Quotient（AQ) score | baseline, after 4,12 weeks of treatment, after 90 days of onset.
Change in Barthel Index score and proportion of subjects with Barthel Index score ≥90 | baseline, after 4,12 weeks of treatment, after 90 days of onset.
Change in the Upper Extremity Fugl-Meyer score | baseline, after 4,12 weeks of treatment, after 90 days of onset.
Change in the total Fugl-Meyer motor score | baseline, after 4,12 weeks of treatment, after 90 days of onset.
Change in the syndrome score of Qi Deficiency and Blood Stasis | baseline, after 4,12 weeks of treatment, after 90 days of onset.
the incidence of New-onset cardiovascular events | during the 20-weeks
Changes in plasma glucose and lipid concentrations and blood coagulate | baseline and after 12 weeks of treatment
physical examination、 laboratory tests and ECG | baseline and after 12 weeks of treatment
the incidence of adverse events | during the 20-weeks
all cause mortality | during the 20-weeks

OTHER OUTCOMES:
The modified Rankin Scale(mRS) score | baseline
the National Health Interview Surveys (NHISS) score | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Wang, Ph.D., Study Director — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences; Yingzhen Xie, M.D., Principal Investigator — Dongzhimen Hospital, Beijing
Locations (13):
- China (13):
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - Langfang TCM Hospital, Langfang, Hebei
  - Luohe Hospital of Chinese Medicine, Luohe, Henan
  - the First affiliated Hospital of Henan University of TCM, Zhengzhou, Henan
  - the affiliated Hospital to Changchun University of Chinese Medicine, Changchun, Jilin
  - 201 Hospital of People's Liberation Army, Dalian, Liaoning
  - Zhongshan Hospital Dalian University, Dalian, Liaoning
  - Second Hospital affiliated to Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Teaching Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing
  - Guang'anmen Hospital Nan District,China Academy of Chinese Medical Sciences, Beijing
  - First Teaching Hospital of Tianjin University of TCM, Tianjin